CLINICAL TRIAL: NCT04485754
Title: Telemedicine Follow-up for Post-Acute Coronary Syndrome Patients
Brief Title: Telemedicine Follow-up for Post-ACS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TeleFU
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: Telemedicine follow-up visit; Post-ACS rehabilitation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine FU (Experimental): Telemedicine follow-up visit at 1, 3, and 6 months or 1 and 6 months after discharge from hospital.
  Interventions: Other: Telemedicine FU
- Office FU (Active Comparator): Office follow-up visit at 1, 3, and 6 months or 1 and 6 months after discharge from hospital.
  Interventions: Other: Office FU

INTERVENTIONS:
Other: Telemedicine FU — Participant will get telemedicine follow-up visit at 1, 3, and 6 months or 1 and 6 months after discharge from hospital.
  Arms: Telemedicine FU
Other: Office FU — Participant will get office follow-up visit at 1, 3, and 6 months or 1 and 6 months after discharge from hospital.
  Arms: Office FU

SUMMARY:
The aim is to compare the safety of using telemedicine and office visit follow-up in post-acute coronary syndrome patients

DETAILED DESCRIPTION:
Rehabilitation after acute coronary syndrome includes visits to the cardiologist's office at 1, 2, 6 and 12 months after discharge. Due to the Covid-19 pandemic, visiting a cardiologist's office maybe impossible. In such cases telemedicine follow-up visit would be reasonable choice. Taking into account the absence of studies in this area, providing investigation evaluating parameters of safety for both methodics is relevant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 40 years
3. PCI with coronary artery stenting for ACS
4. Angiographic success PCI

Exclusion Criteria:

1. Patients with cancer
2. Severe CHF (EF LV <35% or functional class of heart failure III-IV NYHA)
3. Severe valvular heart disease or Prosthetic heart valves.
4. Severe forms of CKD (GFR<30mL/min)
5. Planned staged revascularization during the next 12 months
6. Planned surgery within the next 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
MACCE | 1 year
  Major adverse cardiac and cerebrovascular events: cardiac death, myocardial infarction, or stroke

SECONDARY OUTCOMES:
High level of MT optimization | 1 year
  High Level of Medical Therapy Optimization is defined as a participant meeting all of the following goals: LDL < 1.4 mmol/L and on any statin, blood pressure < 140/90 mm/Hg (<135/85 mm/Hg for patients with diabetes mellitus), on aspirin or other antiplatelet or anticoagulant, and not smoking. High level of medical therapy optimization is missing if any of the individual goals are missing.
PB < 140/90 mm/Hg (<135/85 mm/Hg for Diabetes) | 1 year
  Blood pressure < 140 mm/Hg (<135/85 mm/Hg for for patients with diabetes mellitus)
LDL < 1.4 mmol/L | 1 year
  Low density lipoprotein< 1.4 mmol/L
Not smoking | 1 year
  Not smoking
Decrease in overweight | 1 year
  Decrease in overweight
Aspirin or other antiplatelet or anticoagulant | 1 year
  Adherence to aspirin or other antiplatelet or anticoagulant
Adherence to prescribed medication | 1 year
  Adherence to prescribed at discharge medication
Hospitalization | 1 year
  Hospitalization for cardiac reasons

CONTACTS AND LOCATIONS:
Overall Officials: Ivan S Bessonov, MD, PhD, Principal Investigator — Tyumen Cardiology Research Center
Locations (1):
- Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen, Russia

IPD SHARING:
Plan to Share IPD: No